CLINICAL TRIAL: NCT03637309
Title: Multi-Media Parent-based Intervention to Promote Dental Hygiene Among Young Children: BeReady2Smile
Acronym: BR2S
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DE027001-01
Record Dates: First submitted 2018-07-19; First posted 2018-08-20 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Dental Caries in Children
MeSH Terms: interventions — Amyloid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BeReady2Smile Video and App (Experimental): This arm will test the feasibility of the BeReady2Smile Video and App to promote dental health of young children with a parent education program.
  Interventions: Behavioral: BeReady2Smile Video and App

INTERVENTIONS:
Behavioral: BeReady2Smile Video and App — BeReady2Smile is a coordinated oral health prevention intervention program that includes video content that features demonstrations/content on encouraging brushing, proper loading of toothbrush, brushing duration and frequency, fluoride myths, and limiting sugar sweetened beverages and milk in baby bottles while in bed. BeReady2Smile will also include a mobile application built within a web-based infrastructure, so parents can participate in multi-media educational activities, develop dental health behavior plans, tailor features and receive feedback from the system on a secure website.

SUMMARY:
This application, BeReady2Smile, will promote dental health behavioral parenting strategies among parents by incorporating a behavioral program for their children. Parents use a multimedia coordinated oral health prevention intervention program to promote dental health targeted at parents of young children attending parenting education classes and families receiving home visiting services through Head Start. Once developed, BeReady2Smile will be field tested for usability and usefulness with a group of parents of young children. Parents will rate the level of support needed, confidence in the system, and ease of use at each stage in the development, initiation, and maintenance of the system.

DETAILED DESCRIPTION:
Approximately one out of three 2- to 5-year-old children in the United States has experienced caries (tooth decay). The American Academy of Pediatric Dentistry and American Academy of Pediatrics provide recommendations for preventive strategies, and recognize that infant, toddler and early childhood oral health is one of the foundations upon which preventive education and dental care must be built to enhance the opportunity for a lifetime free from preventable oral disease. Parents struggle to adopt these preventive strategies at the same time that challenging behaviors emerge in children's psychological development. This combination can make it very difficult to build the foundation of oral health practices that the American Academy of Pediatric Dentistry and American Academy of Pediatrics recommends. There is a strong body of evidence supporting the use of behavioral parenting strategies in dealing with child behavioral problems. The proposed project introduces behavioral parent training strategies in concert with efforts to address other known parental barriers to provide an effective vehicle to promote dental health with a universal prevention intervention.

This private/public collaboration between Oregon Research Behavioral Intervention Strategies, Oregon Research Institute & The Oregon Community Foundation will leverage resources and competencies to create a commercially viable coordinated oral health prevention intervention program to promote dental health targeted at parents of young children attending parenting education classes and families receiving home visiting services through Head Start. The program includes a video that can be shown in parenting education classes to engage parents on oral health and a mobile/web application to drive behavioral change.

In this Phase I application, the investigators propose developing a coordinated oral health prevention intervention program, "BeReady2Smile", including video and mobile/web- application. An initial proof of concept version of this program and reminder set will be developed in the Phase I project and then tested for feasibility/usability among parents of young children. BeReady2Smile will include video content that features demonstrations/content on encouraging brushing, proper loading of toothbrush, brushing duration and frequency, fluoride myths, and limiting sugar sweetened beverages and milk in baby bottles while in bed. BeReady2Smile will also include a mobile application built within a web-based infrastructure, so parents can participate in multi-media educational activities, develop dental health behavior plans, tailor features and receive feedback from the system on a secure website. The long-term goal of BeReady2Smile is to help parents provide the foundation for a lifetime free from preventable oral disease.

ELIGIBILITY:
Inclusion Criteria:

* Adults attending parent support groups with children 0-6 years.

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-09-08 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Satisfaction with BeReady2Smile | Up to 16 weeks
  Satisfaction was assessed by participants' ratings on a 1-4 scale (from "Liked very much" to "Not at all liked") of the question "How much did you like BeReady2Smile for learning the information taught?"

SECONDARY OUTCOMES:
Attitudes toward Dental Behaviors: Importance and Intention to Brush Child's Teeth | Baseline, up to 16 weeks
  Parental attitudes toward dental behaviors were assessed by four scales included in the questionnaires developed by Adair and colleagues (2004) including the 'Importance and Intention to Brush Child's Teeth' (five items). Response options range from 'strongly agree' (=1) to 'strongly disagree' (=5).
Attitudes toward Dental Behaviors: Parental Efficacy in Relation to Child Toothbrushing | Baseline, up to 16 weeks
  Parental attitudes toward dental behaviors were assessed by four scales included in the questionnaires developed by Adair and colleagues (2004) that included Parental Efficacy in Relation to Child Toothbrushing' (six items). Response options range from 'strongly agree' (=1) to 'strongly disagree' (=5).
Attitudes toward Dental Behaviors: Perceived Seriousness of Tooth Decay in Children | Baseline, up to 16 weeks
  Parental attitudes toward dental behaviors were assessed by four scales included in the questionnaires developed by Adair and colleagues (2004) that included Perceived Seriousness of Tooth Decay in Children' (seven items). Response options range from 'strongly agree' (=1) to 'strongly disagree' (=5).
Attitudes toward Dental Behaviors: Chance Control - Decay Occurs by Chance | Baseline, up to 16 weeks
  Parental attitudes toward dental behaviors were assessed by four scales included in the questionnaires developed by Adair and colleagues (2004) that includes 'Chance Control - Decay Occurs by Chance' (five items). Response options range from 'strongly agree' (=1) to 'strongly disagree' (=5).
Application Usage | up to 16 weeks
  Activity logs tracked the use of the BeReady2Smile website with a time and date for every online activity.

CONTACTS AND LOCATIONS:
Overall Officials: David R Smith, PhD, Principal Investigator — Orbis
Locations (1):
- Oregon Research Institute, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided